CLINICAL TRIAL: NCT00957619
Title: Study of the Protective Effect of Mechanism of Pentoxyfilline After Major Liver Resection Under Inflow Occlusion (Pringle Manoeuvre)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ksenija Slankamenac, MD PhD, University of Zurich
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: StV 7-2006
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Liver Regeneration
Keywords: pentoxyfilline; liver regeneration; major liver resection; reduction of the I/R injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pentoxyfilline group (Active Comparator): pentoxyfilline group
  Interventions: Drug: pentoxyfilline
- placebo group (Placebo Comparator): placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pentoxyfilline — The total dose of 1 mg/kg/h will be used. At the preoperative day half of the daily dose will be given as a 4-hour short-term infusion within 24 hours before surgery. Afterwards, a continuous intravenous infusion of PTX 1 mg/kg of body weight per hour will be started intra-operatively and will be continued for a total of 72 hours after surgery.
  Arms: pentoxyfilline group
Drug: Placebo — This group will be treated with saline solution at the same time points. The infusion volume and infusion rate of saline solution correspond to that of the PTF group.
  Arms: placebo group

SUMMARY:
The investigators hypothecate that pentoxyfilline increase significantly the liver regeneration and reduces significantly ischemia and reperfusion (I/R) injury in major liver using aspartate aminotransferase (AST) and alanine aminotransferase (ALT) as marker of I/R injury.

DETAILED DESCRIPTION:
Liver resection is for many patients with primary or secondary hepatic malignancies the only curative treatment option. Often, the complete clearance of the hepatic tumor disease can be only achieved by extended liver resections. Clinical studies have demonstrated that intra-operative blood loss is associated reduced outcome after major liver resection. An effective strategy to reduce blood loss is the occlusion of the portal triad (Pringle manoeuvre). On the other hand, inflow occlusion results in ischemia- and reperfusion (I/R) injury. Randomized trials have shown that ischemic preconditioning (10 min clamping, 10 min reperfusion) and intermittent clamping (15 min clamping, 5 min reperfusion) result in reduction of the I/R injury. Another potential strategy to reduce I/R injury is the pharmacological protection. One promising drug is pentoxyfilline (PTF) which has vasodilative and hemorheologic effects. Furthermore, PTF suppresses the TNF release. These effects may be also protective in major liver resection under inflow occlusion (Pringle manoeuvre)and increase the liver regeneration. Therefore, we designed a randomised prospective trial to investigate the effects of PTF treatment in liver resection under inflow occlusion. The specific aims of the research project are:The investigators hypothecate that pentoxyfilline increases significantly the liver regeneration and reduces significantly ischemia and reperfusion (I/R) injury in liver using aspartate aminotransferase (AST) and alanine aminotransferase (ALT) as marker of I/R injury.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Major liver resection (hemihepatectomies and extended hemihepatectomies) for benign and malignant lesions
* Macroscopic and microscopic normal liver parenchyma
* No underlying liver disease
* Normal preoperative liver tests (quick, bilirubin, AST, ALT)
* Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Minor liver resections (less than hemihepatectomies) or wedge resections
* Macroscopic and microscopic appearance of liver fibrosis or cirrhosis
* Underlying liver disease such as viral hepatitis, cirrhosis, etc.
* Pathological preoperative liver tests (quick, bilirubin, AST, ALT)
* Intolerance to xanthine derivatives
* History of myocardial or cerebrovascular insult
* Total vascular exclusion during liver resection
* Intra-operative detection of unresectable tumor disease
* No signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
I. To determine the regeneration of the liver after liver resection with and without PTF treatment | pre- and up to day 8 after liver resection

SECONDARY OUTCOMES:
Il-6, TNF, procalcitonin for regeneration.AST & ALT peak for ischemic reperfusion injury. If PTF treatment has protective effects in steatotic/fibrotic liver. | pre- and up to 8 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain Clavien, MD, PhD, Principal Investigator — Departmente of Visceral and Transplantation Surgery
Locations (1):
- University Hospital Zurich, Department of Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland